CLINICAL TRIAL: NCT01000051
Title: Eltrombopag for Post Transplant Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0106; NCI-2011-01099 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Thrombocytopenia
Keywords: Transplant Thrombocytopenia; Hematopoietic cell transplantation; HCT; Low platelet count; Bleeding; Blood clot; Stem Cell Transplant; Blood And Marrow Transplantation; Eltrombopag; Promacta
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage; Thrombosis | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Experimental): Starting dose 50 mg/day orally for 8 weeks
  Interventions: Drug: Eltrombopag
- Placebo (Placebo Comparator): Once a day orally for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Starting daily dose 50 mg orally on empty stomach (1 hour before or 2 hours after a meal) for 8 weeks. East Asians start at 25 mg daily.
  Other Names: Promacta
  Arms: Eltrombopag
Drug: Placebo — Once a day, orally for 8 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if eltrombopag can help to improve platelet counts in patients with low platelets after they have had a stem cell transplant. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Platelets are cells that help the blood clot. Platelet counts are often lower after receiving a stem cell transplant. When the number of platelets in your body gets too low, it can cause bleeding. Eltrombopag is designed to imitate a protein in your body that helps make platelets. This may help your platelet counts stay normal.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups:

* If you are in Group 1, you will receive eltrombopag.
* If you are in Group 2, you will receive a placebo. A placebo is a substance that looks like the study drug but has no active ingredients.

If you are 1 of the first 20 participants enrolled in this study, you will have an equal chance of being assigned to either group. If you join the study after 20 participants have been enrolled, you will have a better chance of being assigned to Group 1 if eltrombopag has been shown to be more effective.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take the study drug/placebo pills by mouth 1 time each day while you are on study. The study drug/placebo should be taken on an empty stomach (1 hour before or 2 hours after food/drink). You may drink water, coffee, and/or tea with the study drug/placebo. You should drink any coffee or tea without milk or cream.

The dose of study drug/placebo may be adjusted (raised or lowered) throughout the study based on your reaction to the study drug/placebo.

Study Visits:

Every 2 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any side effects you may have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for PK testing.
* Blood (about 1 tablespoon) will be drawn to check your immune system.

If your blood tests show that you may have fiber deposits (build-up) in the bone marrow, you will have a bone marrow biopsy to check the status of the disease

If you have symptoms of cataracts (clouding of the lens of the eye) anytime during the study, you will have an eye exam.

Length of Study:

You will take the study drug for up to 8 weeks. You will have study visits for 12 weeks. You will be taken off study if you have intolerable side effects.

End-of-Treatment Visit:

After completion of study drug, you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any side effects you may have had.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* Blood (about 1 tablespoon) will be drawn to check your blood's clotting ability.
* Blood (about 1 tablespoon) will be drawn to check your immune system.

Weeks 10 and 12 (+/- 3 days), you will have the following tests and procedures performed:

* You will have a telephone interview.
* You will be asked about any side effects you may have had.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* Blood (about 1 tablespoon) will be drawn to check your blood's clotting ability.
* You will either have blood drawn locally or where you live regionally.

Within the 3 months after your last dose of study drug, you will have a bone marrow biopsy to check the status of the disease and an eye exam. The eye exam may be performed sooner if you develop symptoms of a cataract, such as blurry vision.

This is an investigational study. Eltrombopag is FDA approved and commercially available for the treatment of low platelet counts in patients with idiopathic thrombocytopenic purpura (ITP -- a severe bleeding disease). Its use in patients with low platelet counts after a stem cell transplant is investigational.

Up to 64 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/= 35 days post HCT with Platelet count </= 20 x 10^9/l sustained for 7 days or patients are platelet transfusion dependent, and
2. Neutrophil count >/= 1.5 x 10^9/l anytime within the last seven days before enrollment. Patients can be on myeloid or erythroid growth factors for example filgrastim), and
3. Age >/= 18

Exclusion Criteria:

1. Recurrence or progression of primary malignancy after HCT
2. ALT >/= 2.5 times the ULN
3. Serum bilirubin >2mg/dl (unless due to Gilbert's syndrome)
4. Documented deep vein thrombosis within 1 year before enrollment on the study, except if upper arm thrombosis related to central venous catheters, within 3 months before enrollment on the study.
5. ECOG Performance status >2
6. Pregnancy: Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. A woman of child-bearing potential is defined as a woman who has not been naturally post-menopausal for at least 12 consecutive months or with no previous surgical sterilization. A negative pregnancy test result will be required before any study drug is given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02-17 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants that was enrolled was taken off the study before the randomization process, therefore not included in the participants that started.
Period: Overall Study
Arm/Group | Eltrombopag | Placebo
Started | 42 | 18
Completed | 39 | 17
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Disease Progression | 1 | 0
Not completed — Serious noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag | Placebo | Total
Number analyzed (Participants) | 39 | 17 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 14 | 51
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 23
  Male | 22 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 33 | 13 | 46
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 28 | 14 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Efficacy of Eltrombopaq and Placebo
Description: Comparison of the efficacy of eltrombopag and placebo in patients with thrombocytopenia post hematopoietic cell transplantation (HCT).
Time Frame: Baseline to Day 57
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 39 | 17
Participants
  Achieved platelet count >/= 30 x 10 | 15 | 5
  Achieved platelet count >/= 50 x 10 | 9 | 0
  Platelet count < 30x 10 | 15 | 12

ADVERSE EVENTS:
Time Frame: Through study completion, average of 12 weeks
Arm/Group | Eltrombopag | Placebo
All-Cause Mortality (participants affected / at risk) | 5/39 | 4/17
Serious Adverse Events (participants affected / at risk) | 14/39 | 3/17
Other Adverse Events (participants affected / at risk) | 31/39 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=39) | Placebo (N=17)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 3 | 0
Ataxia (Blood and lymphatic system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
GI graft vs host disease (Gastrointestinal disorders) | 1 | 0
Death/Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections (Infections and infestations) | 5 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=39) | Placebo (N=17)
Creatinine increased (Renal and urinary disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 12 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 5
Vomitting (Gastrointestinal disorders) | 3 | 3
Alanine aminotransferanse increased (Hepatobiliary disorders) | 3 | 6
Ascites (Hepatobiliary disorders) | 1 | 0
Aspatate aminotransferase increased (Hepatobiliary disorders) | 1 | 1
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 3 | 4
Hemorrhage/Urinary Tract (Renal and urinary disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Infection (Infections and infestations) | 7 | 6
Petechiae (Blood and lymphatic system disorders) | 1 | 3
Bilirubin increased (Hepatobiliary disorders) | 10 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT01000051/Prot_SAP_000.pdf